CLINICAL TRIAL: NCT00103727
Title: A Multicenter, Double-Blind, Double-Dummy, Placebo-Controlled, Randomized, Parallel Group Evaluation of the Efficacy and Safety of a Fixed-Dose of Talnetant Versus Placebo Versus Risperidone in Subjects With Schizophrenia
Brief Title: Study Of Talnetant Versus Placebo And Risperidone In Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB-223412/093
Record Dates: First submitted 2005-02-14; First posted 2005-02-15 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Schizophrenia
Keywords: paranoid; catatonic; undifferentiated types; disorganized
MeSH Terms: conditions — Schizophrenia; Catatonia | interventions — SB 223412; Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- talnetant (Experimental): 200mg, 400mg, 600mg) twice a day
  Interventions: Drug: Talnetant
- placebo (Placebo Comparator): placebo
  Interventions: Other: placebo
- risperidone (Active Comparator): 3mg twice a day
  Interventions: Other: risperidone

INTERVENTIONS:
Drug: Talnetant — talnetant
  Arms: talnetant
Other: placebo — Placebo Comparator
  Arms: placebo
Other: risperidone — Active Comparator
  Arms: risperidone

SUMMARY:
This study will evaluate whether talnetant (200mg, 400mg, 600mg) twice a day is effective compared to placebo and risperidone 1-3mg twice a day in treating the positive and negative symptoms of schizophrenia. Study subjects will be treated with study drug for up to 6 weeks and will then return for a follow-up visit 2 weeks later. About 275 patients with schizophrenia will be enrolled in this study.

ELIGIBILITY:
Inclusion criteria:

* Subjects must have schizophrenia which is not secondary to another medical condition or substance abuse.
* Require inpatient hospitalization.
* Woman may enroll only if they are not of child-bearing potential OR are on a protocol-approved birth control method.

Exclusion criteria:

* Subject is in their first episode of schizophrenia.
* Subject has other psychotic disorders or bipolar disorder.
* Subject has schizophrenia symptoms from taking another medicine or drug of abuse, or due to a general medical condition.
* Subject has a recent history of substance dependence/dependence, or tests positive for illicit drug.
* Subject has an unstable medical disorder, or any significant medical disorder including autistic disorder, organic brain disease, liver dysfunction, epilepsy or seizures, or is at increased risk of developing cerebrovascular problems like stroke.
* Subject has any significant abnormalities in any of the screening tests (ECGs, labs, physical examinations, etc.).
* Subject poses a current serious suicidal or homicidal risk.
* Subject has a positive pregnancy test, or is lactating or planning to become pregnant within one month of the study.
* Subject has recently or is currently participating in another clinical study.
* Subject is stabilized on their current schizophrenia treatment.
* Subject needs to take any of the medicines not permitted in the study, or has recently had ECT (electroconvulsive therapy) or TMS (transcranial magnetic stimulation).
* Subject was non-responsive to two or more adequate trials of antipsychotic treatments over the past 2 years.
* Subject has had an allergic or significant reaction to any of the study drugs, or can't take risperidone.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2004-12; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is change in the Positive and Negative Syndrome Scale (PANSS) at Week 6 compared to baseline values. | 6 weeks

SECONDARY OUTCOMES:
The secondary measures assess both efficacy (cognition, depression) as well as a variety of safety/tolerability endpoints (adverse events, motor function, laboratory measures). | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- United States (21):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Cerritos, California
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, Glendale, California
  - GSK Investigational Site, National City, California
  - GSK Investigational Site, Oceanside, California
  - GSK Investigational Site, Pico Rivera, California
  - GSK Investigational Site, Rosemead, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Oak Brook, Illinois
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Clementon, New Jersey
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Irving, Texas
  - GSK Investigational Site, Richmond, Virginia